CLINICAL TRIAL: NCT03472469
Title: MAST Trial: Multi-modal Analgesic Strategies in Trauma
Acronym: MAST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, John Andrew Harvin, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-18-0036; KL2TR000370 (NIH); UL1TR000371 (NIH)
Record Dates: First submitted 2018-03-13; First posted 2018-03-21 (Actual); Results first posted 2021-06-10 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Nonspecific Pain Post Traumatic Injury
MeSH Terms: interventions — Ketorolac; Celecoxib; Naproxen; Tramadol; Pregabalin; Gabapentin; Lidocaine; Analgesics, Opioid; Anesthesia, Conduction

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Original MMPR - descending dose arm (Active Comparator): Drugs are scheduled around the clock as follows: 1. Acetaminophen 1g intravenously (IV)/per oral (PO) q6 hours in the first 48 hours, and Acetaminophen 1g PO q6 hours thereafter; 2. Ketorolac 30mg IV once and Celebrex 200mg PO q12 hours in the first 48 hours, and Naproxen 500mg PO q12 hours thereafter; 3. Tramadol 100mg PO q6 hours in the first 48 hours, and Tramadol 100mg PO q6 hours thereafter; 4. Pregabalin 100mg PO q8 hours in the first 48 hours, and Gabapentin 300mg PO q8 hours thereafter; 5. Lidocaine patch q12 hours in the first 48 hours, and Lidocaine patch q12 hours thereafter; and 6. Opioids (Regional anesthesia) in the first 48 hours, and Opioids and Regional anesthesia thereafter.
  Interventions: Drug: Acetaminophen IV/PO; Drug: Acetaminophen PO; Drug: Ketorolac; Drug: Celebrex; Drug: Naproxen; Drug: Tramadol; Drug: Pregabalin; Drug: Gabapentin; Drug: Lidocaine; Drug: Opioids; Drug: Regional anesthesia
- MAST MMPR - escalating dose arm (Active Comparator): Drugs are scheduled around the clock as follows: 1. Acetaminophen 1g PO q6 hours at admission and thereafter; 2. Ketorolac 30mg IV once and Naproxen 500mg PO q12 hours at admission and thereafter; 3. No drug; 4; Gabapentin 300mg PO q8 hours at admission and thereafter; 5. Lidocaine patch q12 hours at admission and thereafter; and 6. Tramadol and Opioids and Regional anesthesia at admission and thereafter.
  Interventions: Drug: Acetaminophen PO; Drug: Ketorolac; Drug: Naproxen; Drug: Gabapentin; Drug: Lidocaine; Drug: Opioids; Drug: Regional anesthesia

INTERVENTIONS:
Drug: Acetaminophen IV/PO — Acetaminophen 1g IV/PO every 6 hours
  Arms: Original MMPR - descending dose arm
Drug: Acetaminophen PO — Acetaminophen 1g PO every 6 hours
Drug: Ketorolac — Ketorolac 30mg IV once
Drug: Celebrex — Celebrex 200mg PO every 12 hours
  Arms: Original MMPR - descending dose arm
Drug: Naproxen — Naproxen 500mg PO every 12 hours
Drug: Tramadol — Tramadol 100mg PO every 6 hours
  Arms: Original MMPR - descending dose arm
Drug: Pregabalin — Pregabalin 100mg PO every 8 hours
  Arms: Original MMPR - descending dose arm
Drug: Gabapentin — Gabapentin 300mg PO every 8 hours
Drug: Lidocaine — Lidocaine patch every 12 hours
Drug: Opioids — Opioid options include: Oral Opioids (Codeine, Tramadol, Hydrocodone, Oxycodone, Methadone, Morphine, Hydromorphone); Transdermal Opioid (Fentanyl); Intravenous Opioids (Morphine, Hydromorphone, Fentanyl)
Drug: Regional anesthesia — Regional anesthesia

SUMMARY:
This is a comparative effectiveness study of current pain management strategies in acutely injured trauma patients. Two different multi-modal, opioid minimizing analgesic strategies will be compared [original multimodal pain regimen (MMPR) compared to multi-modal analgesic strategies for trauma (MAST) MMPR].

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the trauma service who are 16 years and older.

Exclusion Criteria:

* pregnant
* prisoner
* patients placed in observation (i.e. not admitted to the hospital)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1561 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2019-07-03 (Actual); Study Completion 2019-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Harvin, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harvin JA, Green CE, Vincent LE, Motley KL, Podbielski J, Miller CC, Tyson JE, Holcomb JB, Wade CE, Kao LS. Multi-modal Analgesic Strategies for Trauma (MAST): protocol for a pragmatic randomized trial. Trauma Surg Acute Care Open. 2018 Aug 19;3(1):e000192. doi: 10.1136/tsaco-2018-000192. eCollection 2018. PMID 30206549
- [Result] Harvin JA, Albarado R, Truong VTT, Green C, Tyson JE, Pedroza C, Wade CE, Kao LS; MAST Study Group. Multi-Modal Analgesic Strategy for Trauma: A Pragmatic Randomized Clinical Trial. J Am Coll Surg. 2021 Mar;232(3):241-251.e3. doi: 10.1016/j.jamcollsurg.2020.12.014. Epub 2021 Jan 21. PMID 33486130

RESULTS

PARTICIPANT FLOW:
Groups:
- MAST MMPR - Escalating Dose Arm: Drugs are scheduled around the clock as follows: 1. Acetaminophen 1g intravenously Drugs are scheduled around the clock as follows: 1. Acetaminophen 1g PO q6 hours at admission and thereafter; 2. Ketorolac 30mg IV once and Naproxen 500mg PO q12 hours at admission and thereafter; 3. No drug; 4; Gabapentin 300mg PO q8 hours at admission and thereafter; 5. Lidocaine patch q12 hours at admission and thereafter; and 6. Tramadol and Opioids and Regional anesthesia at admission and thereafter.
Period: Overall Study
Arm/Group | Original MMPR - Descending Dose Arm | MAST MMPR - Escalating Dose Arm
Started | 787 | 774
Completed | 787 | 774
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Original MMPR - Descending Dose Arm | MAST MMPR - Escalating Dose Arm | Total
Number analyzed (Participants) | 787 | 774 | 1561
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 44 [29 to 63] | 45 [28 to 62] | 45 [28 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 248 | 252 | 500
  Male | 539 | 522 | 1061
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 140 | 167 | 307
  Hispanic | 264 | 223 | 487
  Other | 20 | 21 | 41
  White | 363 | 363 | 726
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 787 | 774 | 1561
Number of Participants with Prior Opioid Use [Count of Participants; unit: Participants]
  No | 690 | 685 | 1375
  Yes | 65 | 52 | 117
  Unknown | 32 | 37 | 69
Number of Participants with a History of Smoking [Count of Participants; unit: Participants]
  No | 520 | 524 | 1044
  Yes | 243 | 217 | 460
  Unknown | 24 | 33 | 57
Number of Participants with a Positive Alcohol Screen [Count of Participants; unit: Participants]
  No | 459 | 474 | 933
  Yes | 118 | 130 | 248
  Not performed | 210 | 170 | 380
Number of Participants with a Positive Drug Screen [Count of Participants; unit: Participants]
  No | 319 | 316 | 635
  Yes | 175 | 202 | 377
  Not performed | 293 | 256 | 549
Score on Abbreviated Injury Scale (AIS) - Head [Median (Inter-Quartile Range); unit: units on a scale] — The AIS classifies individual injuries by body region as follows: 0 = No Injury; 1 = Minor; 2 = Moderate; 3 = Serious; 4 = Severe; 5 = Critical; 6 = Maximal (currently untreatable)
  units on a scale | 0 [0 to 2] | 0 [0 to 2] | 0 [0 to 2]
Score on Abbreviated Injury Scale (AIS) - Chest [Median (Inter-Quartile Range); unit: units on a scale] — The AIS classifies individual injuries by body region as follows: 0 = No Injury; 1 = Minor; 2 = Moderate; 3 = Serious; 4 = Severe; 5 = Critical; 6 = Maximal (currently untreatable)
  units on a scale | 2 [0 to 3] | 2 [0 to 3] | 2 [0 to 3]
Score on Abbreviated Injury Scale (AIS) - Abdomen [Median (Inter-Quartile Range); unit: units on a scale] — The AIS classifies individual injuries by body region as follows: 0 = No Injury; 1 = Minor; 2 = Moderate; 3 = Serious; 4 = Severe; 5 = Critical; 6 = Maximal (currently untreatable)
  units on a scale | 0 [0 to 2] | 0 [0 to 2] | 0 [0 to 2]
Injury Severity Score (ISS) [Median (Inter-Quartile Range); unit: units on a scale] — The Injury Severity Score (ISS) assesses the combined effects of injuries in multiple anatomical locations and ranges from from 1 to 75, with 75 being the most severe.
  units on a scale | 14 [9 to 22] | 14 [9 to 22] | 14 [9 to 22]
Number of participants with rib fractures [Count of Participants; unit: Participants] | 364 | 356 | 720
Number of rib fractures [Median (Inter-Quartile Range); unit: rib fractures] | 0 [0 to 4] | 0 [0 to 4] | 0 [0 to 4]
Number of participants with flail segment [Count of Participants; unit: Participants] — Flail segment is the condition of having three or more contiguous ribs fractured in two or more places
  Participants | 47 | 57 | 104
Number of participants with long bone fracture [Count of Participants; unit: Participants] | 252 | 249 | 501
Number of participants with vertebral body fracture [Count of Participants; unit: Participants] | 136 | 144 | 280
Number of participants with pelvis or acetabulum fracture [Count of Participants; unit: Participants] | 142 | 143 | 285
Number of participants with traumatic brain injury [Count of Participants; unit: Participants] | 158 | 147 | 305
Unit of admission [Count of Participants; unit: Participants]
  Floor | 305 | 280 | 585
  Intermediate unit | 186 | 194 | 380
  Intensive care unit | 273 | 279 | 552
  Other | 23 | 21 | 44
Number of participants who underwent laparotomy procedure [Count of Participants; unit: Participants] | 96 | 86 | 182
Number of participants who underwent thoracotomy procedure [Count of Participants; unit: Participants] | 35 | 29 | 64
Number of participants who underwent amputation procedure [Count of Participants; unit: Participants] | 9 | 12 | 21

OUTCOME MEASURES:

1. Primary Outcome: Opioid Use Per Day
Description: Opioid use per day is calculated by tallying the dose equivalency of all opioids received and dividing by the number of days hospitalized. Morphine milligram equivalents (MME) per day are reported.
Time Frame: until discharge from hospital or 30 days post admission (whichever is sooner)
Measure: Median (Inter-Quartile Range); unit: MME per day
Arm/Group | Original MMPR - Descending Dose Arm | MAST MMPR - Escalating Dose Arm
Number analyzed (Participants) | 787 | 774
MME per day | 48 [22 to 74] | 34 [15 to 61]

2. Secondary Outcome: Pain as Assessed by Score on the Numeric Rating Scale (NRS)
Description: An average will be calculated of the daily numeric rating scale (NRS) for pain (0=no pain, 10=worst pain). This assessment is used in verbal participants.
Time Frame: until discharge from hospital or 30 days post admission (whichever is sooner)
Population: This data was only collected from 739 in the Original MMPR arm and 735 in the MAST MMPR arm.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Original MMPR - Descending Dose Arm | MAST MMPR - Escalating Dose Arm
Number analyzed (Participants) | 739 | 735
units on a scale | 3.3 [1.8 to 4.8] | 3.3 [1.8 to 4.7]

3. Secondary Outcome: Pain as Assessed by Score on the Behavioral Pain Scale (BPS)
Description: An average will be calculated of the daily score on the Behavioral Pain Scale (BPS). BPS score ranges from 3-12, with higher scores indicating worse pain. This assessment is used in non-verbal participants.
Time Frame: until discharge from hospital or 30 days post admission (whichever is sooner)
Population: This data was only collected from 156 in the Original MMPR arm and 150 in the MAST MMPR arm.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Original MMPR - Descending Dose Arm | MAST MMPR - Escalating Dose Arm
Number analyzed (Participants) | 156 | 150
score on a scale | 2.5 [2.1 to 3.0] | 2.3 [1.8 to 3.0]

4. Secondary Outcome: Number of Participants Discharged From the Hospital With an Opioid Prescription
Time Frame: Up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Original MMPR - Descending Dose Arm | MAST MMPR - Escalating Dose Arm
Number analyzed (Participants) | 787 | 774
Participants | 527 | 476

5. Secondary Outcome: Number of Participants With Any Opioid-related Complications
Description: Opioid-related complications include ileus, aspiration, unplanned intubation, unplanned admission to an intensive care unit, and use of an opioid-reversal agent.
Time Frame: until discharge from hospital or 30 days post admission (whichever is sooner)
Measure: Count of Participants; unit: Participants
Arm/Group | Original MMPR - Descending Dose Arm | MAST MMPR - Escalating Dose Arm
Number analyzed (Participants) | 787 | 774
Participants
  Unplanned intubation | 16 | 16
  Unplanned admission to the intensive care unit | 30 | 31
  Cardiac arrest with Cardiopulmonary resuscitation (CPR) | 18 | 13
  Ileus | 41 | 45
  Naloxone reversal | 7 | 6

6. Secondary Outcome: Overall Costs
Description: the costs associated with the overall hospitalization or the first 30 days (whichever is sooner) related to post trauma care and complications incurred.
Time Frame: until discharge from hospital or 30 days post admission (whichever is sooner)
Measure: Median (Inter-Quartile Range); unit: dollars
Arm/Group | Original MMPR - Descending Dose Arm | MAST MMPR - Escalating Dose Arm
Number analyzed (Participants) | 787 | 774
dollars | 20093 [9557 to 42492] | 19561 [10238 to 44795]

7. Secondary Outcome: Pharmacy Costs
Description: The costs of the pain medications given during the specified time period.
Time Frame: until discharge from hospital or 30 days post admission (whichever is sooner)
Measure: Median (Inter-Quartile Range); unit: dollars
Arm/Group | Original MMPR - Descending Dose Arm | MAST MMPR - Escalating Dose Arm
Number analyzed (Participants) | 787 | 774
dollars | 507 [240 to 1098] | 397 [183 to 1044]

8. Secondary Outcome: Number of Ventilator Days
Description: The number of days the patient on a ventilator post injury or up to 30 days (whichever is sooner). Zero-inflated models are presented as estimated marginal means (95% Credible Interval). The data reported as "mean" actually refers to "marginal mean," and the data reported as "95% Confidence Interval" actually refers to a "95% Credible Interval."
Time Frame: 30 days
Measure: Mean (95% Confidence Interval); unit: ventilator days
Arm/Group | Original MMPR - Descending Dose Arm | MAST MMPR - Escalating Dose Arm
Number analyzed (Participants) | 787 | 774
ventilator days | 0.08 [0.03 to 0.18] | 0.06 [0.03 to 0.14]

9. Secondary Outcome: Number of Hospital Days
Description: The number of days the patient was hospitalized post injury or up to 30 days (whichever is sooner). Zero-inflated models are presented as estimated marginal means (95% Credible Interval). The data reported as "mean" actually refers to "marginal mean," and the data reported as "95% Confidence Interval" actually refers to a "95% Credible Interval."
Time Frame: 30 days
Measure: Mean (95% Confidence Interval); unit: hospital days
Arm/Group | Original MMPR - Descending Dose Arm | MAST MMPR - Escalating Dose Arm
Number analyzed (Participants) | 787 | 774
hospital days | 4.97 [4.59 to 5.38] | 5.12 [4.72 to 5.55]

10. Secondary Outcome: Number of Intensive Care Unti (ICU) Days
Description: The number of days the patient was in the ICU post injury or up to 30 days (whichever is sooner). Zero-inflated models are presented as estimated marginal means (95% Credible Interval). The data reported as "mean" actually refers to "marginal mean," and the data reported as "95% Confidence Interval" actually refers to a "95% Credible Interval."
Time Frame: 30 days
Measure: Mean (95% Confidence Interval); unit: ICU days
Arm/Group | Original MMPR - Descending Dose Arm | MAST MMPR - Escalating Dose Arm
Number analyzed (Participants) | 787 | 774
ICU days | 0.21 [0.12 to 0.34] | 0.21 [0.13 to 0.35]

11. Secondary Outcome: Degree to Which Function is Limited by Pain as Assessed by Percent of Predicted Daily Incentive Spirometry Volumes (Which is Based on Ideal Body Weight)
Description: Clinical based pain scores ranging from 0 to 10 will be assessed at regular intervals throughout the hospitalization.
Time Frame: until discharge from hospital or 30 days post admission (whichever is sooner)
Population: These data were not collected.
Arm/Group | Original MMPR - Descending Dose Arm | MAST MMPR - Escalating Dose Arm
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Degree to Which Function is Limited by Pain as Indicated by Number of Participants Who Failed to Work With Physical Therapist Due to Pain
Time Frame: until discharge from hospital or 30 days post admission (whichever is sooner)
Population: These data were not collected.
Arm/Group | Original MMPR - Descending Dose Arm | MAST MMPR - Escalating Dose Arm
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From hospital admission to hospital discharge (about 30 days)
Arm/Group | Original MMPR - Descending Dose Arm | MAST MMPR - Escalating Dose Arm
All-Cause Mortality (participants affected / at risk) | 29/787 | 36/774
Serious Adverse Events (participants affected / at risk) | 29/787 | 36/774
Other Adverse Events (participants affected / at risk) | 0/787 | 0/774
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Original MMPR - Descending Dose Arm (N=787) | MAST MMPR - Escalating Dose Arm (N=774)
Death (General disorders) | 29 (787) | 36 (774)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-02): https://cdn.clinicaltrials.gov/large-docs/69/NCT03472469/Prot_SAP_000.pdf